CLINICAL TRIAL: NCT03587519
Title: Short Versus Long Interval to Ileostomy Reversal After Ileal Pouch Surgery for Ulcerative Colitis
Brief Title: Short Versus Long Interval to Ileostomy Reversal After Ileal Pouch Surgery
Acronym: SLIRPS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Adverse Event
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-0929
Record Dates: First submitted 2018-06-26; First posted 2018-07-16 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Ulcerative Colitis; Ileal Pouch; Ileostomy - Stoma
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early ileostomy closure (Experimental): Early ileostomy closure will be performed 7 to 12 days after with ileal j-pouch anal anastomosis (IPAA) and loop ileostomy (IPAA).
  Interventions: Procedure: Early
- Late ileostomy closure (Active Comparator): Late ileostomy closure will be performed 8 - 12 weeks after IPAA.
  Interventions: Procedure: Late

INTERVENTIONS:
Procedure: Early — Early ileostomy closure
  Arms: Early ileostomy closure
Procedure: Late — Late ileostomy closure
  Arms: Late ileostomy closure

SUMMARY:
In patients with ulcerative or indeterminate colitis who undergo ileal pouch anal anastomosis and diverting loop ileostomy (IPAA) surgery* a short interval to loop ileostomy reversal will result in differences in complications and quality of life compared to a long interval to loop ileostomy reversal.

DETAILED DESCRIPTION:
Aim #1: To compare the Comprehensive Complication Index (CCI), the incidence of postoperative complications, including total number of complications per patient, percent of patients with complications, and total number of ostomy-related complications per patient among IPAA patients who have their ileostomy reversed after a short interval compared to a long interval.

Aim #2: To compare the short vs. long interval groups on measures of health-related quality of life (PROMIS) and IPAA functional outcomes

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consents.
* Man or woman between 18 and 64 years of age.
* Ulcerative colitis (UC) or indeterminate colitis (IC) diagnosed by routine clinical, radiographic, endoscopic, and pathological criteria.
* Patient will be scheduled for non-emergent proctocolectomy or completion proctectomy with ileal j-pouch anal anastomosis (IPAA) and loop ileostomy (IPAA).
* Clinical assessment of patient after IPAA surgery indicates that patient is suitable for early ileostomy reversal

Exclusion Criteria:

* Age < 18 or > 64 years
* Colon or rectal cancer
* Crohn's disease or suspected Crohn's disease
* Prednisone dose > 20 mg per day (or equivalent other steroid dose) within 4 weeks of scheduled IPAA
* Body mass index (BMI) equal to or greater than 40 kg/m2
* Hemodynamic instability (persistent pulse rate < 50 or > 120 bpm, systolic blood pressure < 90 or > 160 mm Hg, uncontrolled cardiac arrhythmia, or active vasopressor drug use)
* Organ transplant recipient (e.g. Liver, Kidney, Pancreas)
* Immunosuppression due to chemotherapy drug use or systemic disease.
* Sepsis
* Renal insufficiency (i.e. serum creatinine ? 2 mg/dl or need for dialysis)
* Therapeutic anticoagulation (e.g. venous thromboembolic disease, prosthetic heart valve)
* Blood Hemoglobin < 8 g/dl
* Serum Albumin < 2.5 g/dl
* Individualized decision by the surgeon to exclude the patient based on sound surgical judgment
* Pregnant patients and female patients who do not satisfy the standard of care requirements of participating centers for an elective surgical procedure.
* Clinical assessment of patient after IPAA surgery indicates that patient is not suitable for early ileostomy reversal
* Participation in another clinical trial within the last 30 days, or simultaneous participation in another clinical trial
* Well-founded doubt about the patient's cooperation.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Comprehensive Complication Index at 6 months after randomization. | 6 months
  The CCI® calculator is an online tool to support the assessment of patients' overall morbidity. The Comprehensive Complication Index (CCI®) is based on the complication grading by Clavien-Dindo Classification and implements every occurred complication after an intervention. The overall morbidity is reflected on a scale from 0 (no complication) to 100 (death).

SECONDARY OUTCOMES:
Total number of postoperative complications per patient | 6 months
  Post-operative complications. For example, surgical site infection, venous thromboembolism, lung or heart-related complications, etc.)
Percent of patients with complications | 1-2 month intervals after randomization through 6 months".
  Percentage of patients with one or more postoperative complication such as surgical site infection, venous thromboembolism, lung or heart-related complications, etc.
Total number of stoma related complications per patient | 1-2 month intervals after randomization through 6 months
  Examples: leakage, pain, retraction, prolapse, bleeding, etc.
Health-related quality of life | Once, at 6 months after ostomy closure surgery
  PROMIS questionnaire. This will be used to assess the study patient's overall health, quality of life, physical health, mental health, social activities, relationships, activities of daily living, emotional health, fatigue level, and pain.
IPAA functional outcomes | Once, at 6 months after ostomy closure surgery
  Daily stools, nightly stools, stool seepage, stool incontinence, anti-peristaltic medication use

CONTACTS AND LOCATIONS:
Overall Officials: Jon Vogel, MD, Principal Investigator — University of Colorado, Denver
Locations (8):
- United States (8):
  - Cedars Sinai, Los Angeles, California
  - University of Colorado Denver, Aurora, Colorado
  - Northwestern University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Beth Israel, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Cleveland Clinic, Cleveland, Ohio

REFERENCES:
- [Derived] Vogel JD, Fleshner PR, Holubar SD, Poylin VY, Regenbogen SE, Chapman BC, Messaris E, Mutch MG, Hyman NH. High Complication Rate After Early Ileostomy Closure: Early Termination of the Short Versus Long Interval to Loop Ileostomy Reversal After Pouch Surgery Randomized Trial. Dis Colon Rectum. 2023 Feb 1;66(2):253-261. doi: 10.1097/DCR.0000000000002427. Epub 2023 Jan 6. PMID 36627253

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-11): https://cdn.clinicaltrials.gov/large-docs/19/NCT03587519/Prot_SAP_000.pdf